CLINICAL TRIAL: NCT03738410
Title: A Multi-Lingual, Culturally-Competent Mobile Health Intervention to Reduce Medical Mistrust, Stigma, and Improve Treatment Adherence Among Women Living With HIV/AIDS (WLWH)
Brief Title: An mHealth Intervention to Improve Outcomes for Women With HIV/AIDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lunthita M. Duthely, Research Associate Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 20170287; 5R34DA057150 (NIH)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: HIV/AIDS
Keywords: mHealth; mobile applications; culturally-competent; HIV stigma; Resilience
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This is a qualitative/quantitative trial that utilizes a Sequential to Parallel intervention study design model. The initial 15 participants (first 5 each that speak English, Spanish, or Haitain Creole) will participate in the Qualitative arm. These participants may also be eligible to roll over into the quantitative portion of the study and randomized to either the control group or the mHealth Intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Active Comparator): The control arm will receive standard of care.
  Interventions: Other: Standard of Care Treatment
- Mobile Health Messaging Arm (Experimental): The Patient Navigation and Mobile Health Messaging Arm will receive standard of care, as well as patient navigation assistance and the mobile health intervention. The mHealth intervention includes psycho-educational messaging as well.
  Interventions: Behavioral: Mobile Health Messaging application; Other: Standard of Care Treatment
- Focus Group Arm (No Intervention): The results of the focus groups will contribute to the wording and design of the intervention.

INTERVENTIONS:
Behavioral: Mobile Health Messaging application — Mobile messaging sent to participants over a 12-month period.
  Arms: Mobile Health Messaging Arm
Other: Standard of Care Treatment — Standard of care (SOC) is defined as the usual care a licensed health care provider would give patients to treat HIV/AIDS. SOC associated procedures and policies may vary across clinical settings.
  Arms: Control Arm; Mobile Health Messaging Arm

SUMMARY:
The purpose of this study is:

1. To develop a new mobile health (mHealth) system that will send text messages to remind both pregnant and non-pregnant women with HIV to adhere to their treatment plan (like keeping appointments, fillings prescriptions, and taking their medication) and address individual barriers to HIV care (like stigma, medical mistrust and resilience).
2. The intervention will also include patient navigation and motivational interviewing

2) Investigators also want to see if the mHealth system is feasible, easily accepted and if it will impact patient health in a positive way.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV diagnosis as per the clinic standard
* Female >= 18 years old at enrollment
* Currently active or recently returned into care or newly enrolled
* With two or more previously scheduled visits (12 months prior to study enrollment
* in the 12 months prior to enrollment:
* missed one or more visits or
* viral load detectable (>20 mL) or
* not taking prescribed HIV anti-retroviral medications

Exclusion Criteria:

* men
* women who are cognitively impaired or are not able to consent for themselves
* non-working cell phone
* adolescents < 18 years old at enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identify
Enrollment: 80 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Enrollment | Month 12
  The proportion of participants enrolled and proportion of participants declined enrollment or screen failed out of total number of participants approached.
Acceptability of the mHealth application | Month 12
  The proportion of messages opened, which were received

SECONDARY OUTCOMES:
Change in Clinic Attendance | Baseline, Month 12
  Change in attendance to HIV primary care visits within 12 months of randomization
Change in HIV Stigma | Baseline, Month 12
  Change in measured stigma (AIDS-related Stigma Scale) within 12 months of randomization (range 40=strongly disagree to 160=strongly agree).
Change in Medical Mistrust | Baseline, Month 12
  Change in measured medical mistrust (Group-based Medical Mistrust) within 12 months of randomization (range 12=does not agree at all to 60=completely agrees).
Change in Resilience | Baseline, Month 12
  Change in measured resiliency (Connor-Davidson Resiliency Scale) within 12 months of randomization (range 0=not true at all to 100=true nearly all of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Lunthita M Duthely, Ed.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duthely LM, Sanchez-Covarrubias AP, Prabhakar V, Brown MR, Thomas TES, Montgomerie EK, Potter JE. Medical Mistrust and Adherence to Care Among a Heterogeneous Cohort of Women Living with HIV, Followed in a Large, U.S. Safety Net Clinic. Health Equity. 2021 Sep 24;5(1):681-687. doi: 10.1089/heq.2020.0105. eCollection 2021. PMID 34909537
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Duthely LM, Sanchez-Covarrubias AP, Mohamed AB, Potter JE. A Multilingual, Culturally Competent Mobile Health Intervention to Improve Treatment Adherence Among Women Living With HIV: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jun 19;9(6):e17656. doi: 10.2196/17656. PMID 32438338